CLINICAL TRIAL: NCT01253772
Title: Pulse Oximeter Responses to Multiple Levels of Stable Hypoxia in Neonates
Status: Completed | Type: Observational
Sponsor: SterilMed, Inc. (Industry)
Responsible Party: Garrett Ahlborg, SterilMed, Inc.
Other Study IDs: STER01P
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Validate pulse oximeter sensors in neonates by comparing sensor readings to blood samples during cardiac surgery.

DETAILED DESCRIPTION:
Researchers at the University of California, San Francisco have developed methods that permit them to test multiple pulse oximeter sensors on neonates simultaneously during cardiac surgery. During this type of surgery, the arterial oxygen saturation changes over a wide range, providing an ideal arena for the assessment of neonatal pulse oximeter sensors at many levels of oxygen saturation. Several arterial blood gas samples are typically obtained during these procedures. Saturation of each arterial blood sample is determined by direct oximetry in a hemoximeter and this measurement is compared to the reading displayed on the pulse oximeter.

ELIGIBILITY:
Inclusion Criteria:

* Neonatal patient scheduled to undergo cardiac surgery where routine blood draws would be taken
* Understand and provide signed parental/guardian consent

Exclusion Criteria:

* Failure to obtain parental consent
* Patients shown to have an adverse reaction to medical tape/adhesive

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonatal children undergoing complex cardiac surgical procedures.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2010-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
SpO2 Accuracy Verification Study (ARMS) of ≤ 3% | During Analysis - data were collected anywhere from the beginning of surgery until the completion of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Greg Stratmann, MD, Principal Investigator — University of California, San Francisco